CLINICAL TRIAL: NCT04529889
Title: Gestational Diabetes Mellitus and Its Consequences in Mothers and Offsprings
Brief Title: GDM and Its Consequences in Mothers and Offsprings
Acronym: GDMCMO
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Born in Guangzhou Cohort Study, Guangzhou Women and Children's Medical Center
Other Study IDs: 201943701; 81803251 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2020-07-20; First posted 2020-08-28 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Gestational Diabetes Mellitus; Pregnancy Outcome; Neurodevelopment; Immune Development; Childhood Obesity; Host and Microbiome
Keywords: Hyperglycaemia; Maternal health; Children; Cohort
MeSH Terms: conditions — Diabetes, Gestational; Pediatric Obesity; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood and urine. At delivery: cord, cord blood and placenta. During infancy: dry blood spot and blood of children. During childhood: blood and buccal swab of children; blood of mothers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Gestational diabetes mellitus (GDM) is one of the most common disorders which occured during pregnancy. GDM is not only associated with short-term maternal and fetal adverse outcomes, but also related to a wide range of long-term consequences for both mother and child. The GDM and Its Consequences for mothers and offsprings (GDMCMO) aims to establish a cohort to follow both maternal and offsprings'short-term and long-term outcomes, including fetal malformations including congenital heart diseases, birth weight, preterm birth, caesarean section delivery, body growth and neurodevelopment after birth, obesity, type 2 diabetes and impaired insulin sensitivity and secretion, lung health and allergic diseases later in life for offspring, as well as future type 2 diabetes and cardiovascular risk factors for mother after delivery. Biological samples including blood and tissue samples of mothers and children are also collected during pregnancy and after delivery.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is one of the most common disorders which occured during pregnancy. GDM is not only associated with short-term maternal and fetal adverse outcomes, but also related to a wide range of long-term consequences for both mother and child. Although maternal hyperglycemia often become normal shortly after pregnancy, women with GDM have crucially increased risk of development of type 2 diabetes later in life and the mechanisms are not fully understand. Systematic follow-up of the outcomes related to GDM would be ideal to observe the nature progression of GDM to diabetes and could help to develop preventable targets for intervention. The risks of obesity, the metabolic syndrome, and type 2 diabetes in offspring of mothers with GDM significantly increased 1-7 folds than those whose mothers didn't have GDM. The underlying pathogenic mechanisms behind the impaired metabolic risk profile and other diseases in offspring are unknown, but environmental changes including epigenetic changes induced by exposure to maternal hyperglycaemia and genetic factors may play essential roles. The GDM and Its Consequences for mothers and offsprings (GDMCMO) aims to establish a cohort to follow both maternal and offsprings'short-term and long-term outcomes, including fetal malformations including congenital heart diseases, birth weight, preterm birth, caesarean section delivery, body growth and neurodevelopment after birth, obesity, type 2 diabetes and impaired insulin sensitivity and secretion, lung health and allergic diseases later in life for offspring, as well as future type 2 diabetes and cardiovascular risk factors for mother after delivery. Biological samples including blood and tissue samples of mothers and children are also collected during pregnancy and after delivery. We also aim to identify the high-risk population of mother-child pairs who are more likely to develop these adverse consequences, which might help to improve precise intervention and resource saving and provide evidence for preventable targets development.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women diagnosed with gestational diabetes mellitus
2. Pregnant women intended to eventually deliver in Guangzhou Women and Children's Medical Center
3. Permanent residents or families intended to remain in Guangzhou with their child for no less than 3 years

Exclusion Criteria:

1. Women with pre-gestational diabetes mellitus
2. Women with chronic hypertension or kidney disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women diagnosed with gestational diabetes mellitus during pregnancy and their offsrpings
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2038-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of obesity status during childhood and adolescence | At age of 6 months, 1 year, 3 years, 6 years, 12 years and 18 year
  Weight in kilograms and height in meters were measured by nurses in clinic using standard tools. Weight and height will be combined to report BMI in kg/m^2. Childhood obesity is defined as a BMI equal to or larger than the 95th percentile for age by sex based on WHO Child Growth Standards.

SECONDARY OUTCOMES:
Number of participants with adverse pregnancy outcomes | At delivery
  Including abortion, stillbirth, live birth, macrosomia, preterm birth, low birth weight, caesarean section delivery, and birth defects.
Change of type 2 diabetes status in mothers | At 1 year, 3 years , 6 years, 12 years and 18 year after delivery
  Assessed by testing concentrations of maternal blood glucose.
Change of body composition of mothers | At 42 days, 6 months, 1 year, 3 years , 6 years, 12 years and 18 year after delivery
  Assessed body composition using dual-energy X-ray absorptiometry.
Change of depression symptom of mothers | At 1 year, 3 years , 6 years, 12 years and 18 year after delivery
  Using Edinburgh Postnatal Depression Scale and Self-rating Depression Scale to assess maternal depression. Higher score is considered more depressive.
Change of neurodevelopment at early childhood | age of 6 weeks, 6 months, 1 year and 3 years.
  Assessed by Gesell Developmental Schedules and Ages&Stages Questionnaires which include adaptive, gross motor, fine motor, language, and social function domains. Higher intelligence quotient score in each domain is considered a better outcome. Intelligence quotient of Gesell Developmental Schedules being less than 86 or intelligence quotient of Ages&Stages Questionnaires being no more than -2SD under the mean is defined as suspected development retardation.
Change of lung function during childhood and adolescence | At age of 6 years, 12 years and 18 years.
  Zrs, R5, R20, X5, X20, Fres assessed by impulse oscillometry
Change of Allergic diseases status during childhood and adolescence | At age of 1 year, 3 years, 6 years, 12 years and 18 years.
  Eczema, allergic rhinitis, wheeze, and asthma diagnosed by the doctors or assessed by the standardized questionnaires
Change of type 2 diabetes during childhood and adolescence | At age of 6 years, 12 years and 18 years.
  Assessed by testing concentrations of children's blood glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, MD,PhD, Principal Investigator — Guangzhou Women and Children's Medical Center, China
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qiu X, Lu JH, He JR, Lam KH, Shen SY, Guo Y, Kuang YS, Yuan MY, Qiu L, Chen NN, Lu MS, Li WD, Xing YF, Zhou FJ, Bartington S, Cheng KK, Xia HM. The Born in Guangzhou Cohort Study (BIGCS). Eur J Epidemiol. 2017 Apr;32(4):337-346. doi: 10.1007/s10654-017-0239-x. Epub 2017 Mar 20. PMID 28321694
- [Background] Shen S, Lu J, Zhang L, He J, Li W, Chen N, Wen X, Xiao W, Yuan M, Qiu L, Cheng KK, Xia H, Mol BWJ, Qiu X. Single Fasting Plasma Glucose Versus 75-g Oral Glucose-Tolerance Test in Prediction of Adverse Perinatal Outcomes: A Cohort Study. EBioMedicine. 2017 Feb;16:284-291. doi: 10.1016/j.ebiom.2017.01.025. Epub 2017 Jan 18. PMID 28122694
- [Background] Shen SY, Zhang LF, He JR, Lu JH, Chen NN, Xiao WQ, Yuan MY, Xia HM, Lam KBH, Qiu X. Association Between Maternal Hyperglycemia and Composite Maternal-Birth Outcomes. Front Endocrinol (Lausanne). 2018 Dec 11;9:755. doi: 10.3389/fendo.2018.00755. eCollection 2018. PMID 30619087